CLINICAL TRIAL: NCT00001458
Title: Diagnosis and Treatment of Patients With Heart and Vascular Disease (Training Protocol)
Brief Title: Evaluation of Patients With Heart Disease Not Eligible for Research Protocols
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950047; 95-H-0047
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Treatment; Cardiovascular Disease; Cardiovascular Testing; Heart Disease; Muscle Leg Pain; Leg Pain; Circulation; Peripheral Arterial Disease; Intermittent Claudication; Renal Vascular Disease; Uncontrolled Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiovascular: subjects with cardiovascular symptoms or known disease.

SUMMARY:
An important mission of the National Institutes of Health (NIH) is to develop and carry out research studies designed to improve understanding of disease processes and treatments.

Clinical research continues to become more focused on specific diseases and the signs and symptoms of diseases in specific groups of people and patients.

This study is designed to permit inpatient evaluation and care of patients with heart disease who do not qualify to participate in research studies being conducted by the Cardiology Branch of the National Heart, Lung, and Blood Institute (NHLBI). These patients are valuable to the Cardiology Branch of the NHLBI because they help to improve training and experience of its researchers.

DETAILED DESCRIPTION:
An important mission of the NIH is to the conduct of research that elucidates biological mechanisms, pathogenesis and treatment of diseases. Clinical research has evolved into an increasingly narrow focus on specific diseases and disease presentations in select subgroups of patients. It is desirable and consistent with Clinical Center policy, for clinical investigators to maintain exposure to a more broad spectrum of disease and disease presentations than mandated by the clinical research protocols in order to preserve clinical skills of physician and nursing staff, ensure adequate training of clinical research fellows, and stimulate ideas for future clinical research. This protocol permits evaluation and treatment of patients with cardiovascular diseases who do not fulfill eligibility criteria for participation in existing clinical research protocols, but who are of medical interest for the purpose of training professional staff.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with signs or symptoms or risk of cardiovascular disease may participate in this training protocol. The following is a representative list of the types of patient presentations and potential diagnoses eligible for this protocol:

Coronary artery disease with effort or rest angina or inducible myocardial ischemia as determined by noninvasive testing.

Valvular heart disease.

Cardiomyopathies, including restrictive, congestive, and hypertrophic phenotypes.

Peripheral-artery disease of upper or lower extremities, with intermittent pain with activity (e.g. claudication) or limb-threatening ischemia.

Renovascular disease with uncontrolled hypertension, intermittent pulmonary edema, or evidence of ischemic nephropathy.

Congenital heart disease, with communications between chambers or major vessels

Heart surgery patients treated at the Clinical Center prior to closure of the Heart Surgery Branch in 1990

EXCLUSION CRITERIA:

Pregnancy, for those patients who require testing or treatment requiring dobutamine, gadolinium or contrast media or radiation exposure.

Inability of patient, parent or legal guardian to provide informed consent.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects can be self-referred; referred per PCP or other specialist from any community or area of the world.@@@
Sampling Method: Non-Probability Sample
Enrollment: 7829 (Actual)
Dates: Start 1995-01-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
training of staff | 20 years
  staff becomes familiar or proficient in cardiovascular diagnostic studies.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Brofferio, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1995-H-0047.html